CLINICAL TRIAL: NCT02933515
Title: Merging Yoga and Group OT (MY-OT)
Brief Title: Merging Yoga and Group OT (MY-OT) to Improve Balance and Decrease Fall Risk After Stroke
Acronym: MY-OT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Arlene Schmid, Associate Professor, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-3805H
Record Dates: First submitted 2016-01-14; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: yoga; occupational therapy; stroke
MeSH Terms: conditions — Stroke | interventions — Yoga; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga and occupational therapy (Experimental): twice a week for 8 weeks. one hour of group occupational therapy for fall risk factor management and one hour of yoga for balance
  Interventions: Other: yoga and occupational therapy

INTERVENTIONS:
Other: yoga and occupational therapy — group OT addressed fall risk factors, such as risk factors inside and outside and how to best manage them. yoga was delivered in sitting, standing, and floor postures

SUMMARY:
The long-term goal of this project is to advance best practices in occupational therapy (OT) to manage fall risk factors and reduce fall rates in older adults with stroke. To address this long-term goal, this team previously developed and pilot-tested a therapeutic yoga intervention to improve balance, balance self-efficacy, and fear of falling and a group OT intervention to improve the management of fall risk factors and fear of falling. The success of both prior studies supports Merging Yoga and group OT to improve balance, balance self-efficacy, and fall risk factor management. The objectives of this feasibility study are to 1) further develop, standardize, and manualize the MY-OT intervention and 2) assess change in balance, balance self-efficacy, and fall risk factor management.

DETAILED DESCRIPTION:
8 week intervention of yoga plus occupational therapy. The objectives of this feasibility study are to 1) further develop, standardize, and manualize the MY-OT intervention and 2) assess change in balance, balance self-efficacy, and fall risk factor management.

ELIGIBILITY:
Inclusion Criteria:

* stroke >6 months prior
* 59 years or older
* prior fall or Fear of Falling (FoF)
* completed all stroke rehabilitation
* able to stand with or without an assistive device
* impaired balance with a score of <46 on the Berg Balance Scale
* able to speak English
* score >4 out of 6 on the short Mini Mental Status Exam (Callahan, Unverzagt et al., 2002)
* able and willing to attend twice weekly sessions for 8 weeks.

Exclusion Criteria:

* people with life expectancy <9 months;
* inability to attend sessions due to unresolved transportation issues;
* inability or refusal to provide informed consent

Min Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in balance using Berg Balance Scale | 8 weeks
  14 items to assess balance

SECONDARY OUTCOMES:
Change in balance confidence using Activities Balance Confidence Scale | 8 weeks
  assess balance self-efficacy or confidence to maintain balance while doing different actions
Change in falls management behaviors using the Falls Management Behavior Questionnaire | 8 weeks
  assess the knowledge of how to manage and change behaviors associated with falls

IPD SHARING:
Plan to Share IPD: No